CLINICAL TRIAL: NCT00789568
Title: A Phase 1, Randomized, Placebo- and Active-controlled Crossover Study to Evaluate the Effects of Sapropterin Dihydrochloride Oral Administration on QTc Intervals in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate Effects of Sapropterin Dihydrochloride on QTc Intervals in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QTC-001
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2014-08

CONDITIONS: Phenylketonuria
Keywords: Hyperphenylalanemia due to Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sapropterin Dihydrochloride 100mg/kg and placebo Moxifloxacin (Experimental): A single dose of 100mg/kg of Sapropterin Dihydrochloride taken along with placebo Moxifloxacin.
  Interventions: Drug: sapropterin dihydrochloride; Drug: Moxifloxacin placebo
- Sapropterin Dihydrochloride 20mg/kg and placebo Moxifloxacin (Experimental): A single dose of 20mg/kg of Sapropterin Dihydrochloride taken along with a placebo Moxifloxacin.
  Interventions: Drug: sapropterin dihydrochloride; Drug: Moxifloxacin placebo
- Sapropterin Dihydrochloride placebo and Moxifloxacin (Active Comparator): No placebo tablets for Sapropterin Dihydrochloride will be administered, but instead will be apple juice only, taken along with 400mg of Moxifloxacin.
  Interventions: Drug: Moxifloxacin
- Sapropterin Dihydrocholide placebo and Moxifloxacin placebo (Placebo Comparator): No placebo tablets for Sapropterin Dihydrochloride will be administered, but instead will be apple juice only, taken along with placebo of Moxifloxacin.
  Interventions: Drug: Moxifloxacin placebo

INTERVENTIONS:
Drug: sapropterin dihydrochloride — 20 mg/kg and 100 mg/kg
  Other Names: Kuvan
  Arms: Sapropterin Dihydrochloride 100mg/kg and placebo Moxifloxacin; Sapropterin Dihydrochloride 20mg/kg and placebo Moxifloxacin
Drug: Moxifloxacin — Moxifloxacin is included as a positive control to demonstrate the assay sensitivity based on the expected increased QTc response.
  Arms: Sapropterin Dihydrochloride placebo and Moxifloxacin
Drug: Moxifloxacin placebo — Moxifloxacin placebo tablet
  Arms: Sapropterin Dihydrochloride 100mg/kg and placebo Moxifloxacin; Sapropterin Dihydrochloride 20mg/kg and placebo Moxifloxacin; Sapropterin Dihydrocholide placebo and Moxifloxacin placebo

SUMMARY:
Sapropterin dihydrochloride (subsequently referred to as sapropterin) (Kuvan®) was approved by the FDA for the treatment of hyperphenylalaninemia in 2007. Preclinical and clinical studies and post-marketing surveillance have not demonstrated any specific cardiovascular concerns with sapropterin (Kuvan®). Nonetheless, nonantiarrhythmic drugs may have the potential to prolong QT interval, leading to potentially fatal ventricular tachycardias, including torsades de pointes. As part of the post-marketing commitment, a thorough QT/QTc study will be conducted according to ICH guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent, after the nature of the study has been explained, and prior to any research-related procedures.
* Sexually active subjects must be willing to use an acceptable method of contraception (double barrier) while participating in the study from screening onwards and for at least 4 weeks after the last dose of study drug.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
* Willing and able to comply with all study procedures.
* Healthy male and female subjects between 18 and 50 years of age, inclusive.
* Body mass index (BMI) of ≥ 18 to < 30 kg/m2 inclusive.
* Blood pressure in the range of 90 140 mmHg systolic and 50 90 mmHg diastolic at Screening and Check-in. Blood pressures can be repeated up to three times within 10 minutes of initial assessment while remaining in the supine position.
* No clinically significant 12-lead ECG abnormalities; and a QTc interval < 450 ms for males and < 470 ms for females and a resting heart rate between 45 90 beats/minute at Screening and Check-in.

Exclusion Criteria:

* Has known hypersensitivity to sapropterin or its excipients, or moxifloxacin.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Concurrent disease or condition that would interfere with study participation or safety or any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
* History of clinically significant cardiac condition, eg, myocardial ischemia (including angina) or infarction, congestive heart failure, left ventricular hypertrophy, or cardiomyopathy.
* Screening, Check-in, or Baseline ECG shows any of the following:

  * Sinus arrhythmia with unacceptable rate variation as judged by the Investigator.
  * Excessive heart rate variation at rest, in the Investigator's opinion.
  * PR interval > 210 ms.
  * QRS interval > 110 ms.
  * QRS and/or T wave that the Investigator judges to be unfavorable for consistently accurate QT measurements (eg, indistinct QRS onset, low amplitude T wave, inverted or terminally inverted T wave, merged T and U waves, or indistinct T offset, prominent U-wave that affects QT measurement).
* Neuromuscular artifact that cannot be readily eliminated.
* Documented history of arrhythmias (eg, ventricular arrhythmias and atrial fibrillation).
* Clinically significant electrolyte disturbances at Screening or Check-in (eg, hypo or hyperkalemia or hypocalcemia) or any condition that could lead to electrolyte disturbances (eg, eating disorder), in the Investigator's opinion.
* History of palpitations, seizures, unexplained syncopal episodes, or symptomatic arrhythmias.
* History of additional risk factors for torsade de pointes (eg, history of near-drowning survival due to loss of consciousness, family history of long QT syndrome, or family history of unexplained early sudden death).
* Any condition that, in the opinion of the Investigator, may compromise absorption, metabolism, or elimination of moxifloxacin.
* History of cancer within the last five years, with the exception of adequately treated basal cell carcinoma.
* Known allergy or intolerance to any compound in the test products or any other closely related compound, such as any member of the quinolone class of antimicrobial agents.
* Unresolved clinically significant laboratory findings, in the Investigator's opinion.
* Positive antibody screen for HBsAg, hepatitic C virus (HCV), or human immunodeficiency virus (HIV).
* Acute illness or febrile event within 72 hours of Check-in.
* Use of tobacco or nicotine-containing products within the last 30 days or have a positive urine test for cotinine prior to Check-in.
* History of alcohol or drug abuse (according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition [DSM-IV] criteria) within 12 months prior to Check-in or have a positive urine test for alcohol or substances of abuse at Screening or Check-in.
* Use of alcoholic beverages, caffeine, and grapefruit-containing products 72 hours prior to dosing and until completion of study.
* Subjects who have taken:

  * Any prescription medications or over-the-counter medications including herbal products (eg, St. John's Wort, milk thistle), antacids and nonsteroidal anti-inflammatory medication for acute pain for more than 5 days within 30 days (or 5 elimination half-lives, whichever is longer) of commencing study drug dosing, with the exception of hormonal contraceptives (oral, implant, patch or injections), including Depo-Provera®. For drugs with an elimination half-life greater than 10 days, the prohibition of prior use will be extended to 60 days.
  * Any planned concomitant medication while in the study, including antacids that contain calcium, magnesium, or aluminum (eg, Rolaids or Tums), the ulcer medicine sucralfate (Carafate), or vitamin or mineral supplements that contain calcium, iron, or zinc from 48 hours prior to Baseline (Day -1) and until completion of the study.
* Any psychiatric, behavioral, or neuromuscular condition that may compromise the Investigator's evaluation of drug effect.
* History of intentional suicidal ideation, suicide attempts, depression requiring treatment, or significant depression in the opinion of the Investigator.
* Subjects who cannot tolerate a controlled, quiet study environment, including avoidance during specified timepoints of music, TV, movies, games, and activities that may cause excitement, emotional tension, or arousal.
* Subjects who cannot tolerate the study-specified diet.
* Subjects who are unwilling to comply with study rules, including attempting to void at specified times (prior to ECG timepoints) or maintain quiet, motionless supine posture during specified timepoints.
* Rigorous exercise ≤ 72 hours prior to Check-in or subjects who will not agree or be able to refrain from rigorous exercise until completion of study.
* In the opinion of the Investigator, the presence of any other behavior or condition that increases the risk to individual safety or risk of compromising study objectives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine if a single supratherapeutic dose of sapropterin or a single therapeutic dose of sapropterin has an effect on cardiac repolarization compared with placebo as a change from baseline measured by the subject specific QT correction formula(QTci) | Complete study

SECONDARY OUTCOMES:
Determine if there is a pharmacodynamic relationship between the duration of the QT/QTc intervals and the plasma concentration of sapropterin | Complete Study
To obtain additional pharmacokinetic information for oral sapropterin at the proposed therapeutic and supra-therapeutic doses. | Complete Study
To generate additional safety information | Complete Study

CONTACTS AND LOCATIONS:
Overall Officials: Don Nwose, MD, Study Director — BioMarin Pharmaceutical
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States